CLINICAL TRIAL: NCT04984161
Title: The Effect of Stoma Care Education on the Knowledge and Skill Levels of Pediatric Surgery Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ESRA ARDAHAN AKGUL, research assistant, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TUBITAK 2209
Record Dates: First submitted 2021-07-25; First posted 2021-07-30 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Stoma Ileostomy; Stoma Colostomy; Nurse's Role; Pediatric Surgery
Keywords: stoma care; pediatric surgery; nurse
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: education — The aim of this project is to examine the effect of stoma care education on the knowledge and skill levels of pediatric surgery nurses about stoma care.

SUMMARY:
This project; It is a quasi-experimental prospective study in a single group pre-test post-test order. No randomization will be made in the selection of the sample, and 30 nurses working in the Pediatric Surgery Clinic in hospitals in Izmir and meeting the inclusion criteria will be included in the study. The data of the study will be collected through the Nurse Descriptive Characteristics Questionnaire and the Pediatric Stoma Care Knowledge and Skills Questionnaire. Pre-training introductory characteristics and pediatric stoma care knowledge and skill level of all nurses participating in the study will be measured. After the measurement, the nurses participating in the study will be given training on pediatric stoma care. Immediately after the training and three months later, the pediatric stoma care knowledge and skill levels of the nurses participating in the study will be re-measured. The introductory characteristics of the nurses involved in the project will be given as number and percentage distributions. Comparisons between nurses' introductory characteristics and Stoma Knowledge and Skills Questionnaire before and after education; It will be evaluated by non-parametric or parametric appropriate test. Comparisons between nurses' Stoma Knowledge and Skills Questionnaire scores in the pre- and post-education period will be evaluated by non-parametric or parametric appropriate test in dependent groups. The statistical significance value of the project was determined as p≤0.005. It is planned that the results of the project will mediate an international article and statement in which the effect of stoma care education on the knowledge and skill level of pediatric surgery nurses is presented. As a result of the project, if it is determined that stoma care education has an effect on the knowledge and skill level of pediatric surgery nurses, it is predicted that the quality of care of children with stoma who receive care in other institutions and organizations can be increased and the comfort of the child can be increased.

ELIGIBILITY:
Inclusion Criteria:

* Working in the Pediatric Surgery Clinic
* Volunteering to participate in the study

Exclusion Criteria:

-Having received any previous training on stoma care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
nurse's pediatric stoma care skills level | immediately after pediatric stoma care education
  Immediately after pediatric stoma care education, the pediatric stoma care knowledge level of the participating nurses will be measured with the Pediatric Stoma Care Knowledge and Skills questionnaire.
nurse's pediatric stoma care knowledge level | immediately after pediatric stoma care education
  Immediately after pediatric stoma care education, the pediatric stoma care knowledge level of the participating nurses will be measured with the Pediatric Stoma Care Knowledge and Skills questionnaire.
nurse's pediatric stoma care skills level | 3 months after pediatric stoma care education
  3 months after pediatric stoma care education, the pediatric stoma care knowledge level of the participating nurses will be measured with the Pediatric Stoma Care Knowledge and Skills questionnaire.
nurse's pediatric stoma care knowledge level | 3 months after pediatric stoma care education
  3 months after pediatric stoma care education, the pediatric stoma care knowledge level of the participating nurses will be measured with the Pediatric Stoma Care Knowledge and Skills questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Esra ARDAHAN AKGÜL, Study Chair — İzmir Katip Çelebi University
Locations (1):
- Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No